CLINICAL TRIAL: NCT05561595
Title: Transdiagnostic Intervention to Reduce Internalized Health-Related Stigma
Acronym: HEARTS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB202201862; DP2MH132938 (NIH); PRO00041153 (Other: UFIRST)
Record Dates: First submitted 2022-09-27; First posted 2022-09-30 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Obesity; Skin Disease; Cancer; HIV; Diabetes; Chronic Pain
MeSH Terms: conditions — Obesity; Skin Diseases; Neoplasms; Diabetes Mellitus; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healing HEARTS Intervention (Experimental): The Healing Health-Related Stigma (Healing HEARTS) intervention will provide group telehealth sessions adapted from prior disease-specific interventions for internalized stigma and from standard techniques and structures used in evidence-based cognitive-behavioral therapies. Fifty-minute sessions will be delivered weekly for 12 weeks, followed by 2 every-other-week and 2 monthly sessions. Groups will consist of approximately 8-10 participants and will be led by a doctoral- or masters-level clinician in clinical or counseling psychology or social work. Handouts and homework assignments will be used as part of the group meetings. All group sessions will be conducted remotely using telehealth technology.
  Interventions: Behavioral: Healing HEARTS
- Peer Support (Active Comparator): The peer support condition will provide group telehealth sessions without any tailored stigma content. Group sessions will be 50 minutes and will meet weekly for 12 weeks, followed by 2 every-other-week and 2 monthly sessions. Groups will consist of approximately 8-10 participants and will be led by a doctoral- or masters-level clinician in clinical or counseling psychology or social work. All group sessions will be conducted remotely using telehealth technology.
  Interventions: Behavioral: Peer Support
- Waitlist Control (No Intervention): The waitlist control group will not receive any active intervention until after completing week 12 and week 26 assessments. Participants will receive periodical updates and reminders from study staff to enhance retention. After assessments are completed, participants will be provided with 12 weeks of the Healing HEARTS intervention.

INTERVENTIONS:
Behavioral: Healing HEARTS — Session topics will include: psychoeducation; myths and stereotypes; cognitive distortions and restructuring; coping strategies; interpersonal effectiveness; self-efficacy; mindfulness and self-compassion; acceptance and positive self-image; disclosure and finding support; stigma in health care; and empowerment and advocacy.
  Arms: Healing HEARTS Intervention
Behavioral: Peer Support — Peer support groups will cover general topics such as symptom management, stress, and social support. Stigma will not be a formal topic of discussion, and group leaders will be trained to avoid initiating conversations about stigma; however, to capture realistic discussions in peer support groups, participants will not be prohibited from discussing the topic should they bring it up.
  Arms: Peer Support

SUMMARY:
Stigma due to health conditions increases disease burden and adversely impacts health. The internalization of health-related stigma is associated with impaired mental health and quality of life. The current project will test the effects of a novel, transdiagnostic, group counseling intervention, and peer support, to determine the optimal method for helping patients cope with health-related stigma, reducing its internalization, and enhancing patient quality of life.

DETAILED DESCRIPTION:
This randomized controlled trial (RCT) will test in a sample of 195 patients with high levels of internalized health-related stigma the effects of a novel transdiagnostic intervention designed to help patients cope with this stigma and to reduce its internalization. Participants will be randomly assigned to one of three intervention conditions: (1) a group-based counseling intervention designed to target internalized health-related stigma, delivered virtually (i.e., via telehealth); (2) a general peer support group conducted via telehealth without a targeted stigma intervention; or (3) a waitlist control group. The counseling and peer support conditions will provide 12 weekly group sessions, followed by 2 every other week sessions and 2 monthly sessions (16 sessions total over the course of 26 weeks, or 6 months). Participants across all conditions will complete outcome assessment visits at baseline/randomization, week 12, and week 26. The waitlist control group will receive 12 weeks of the group counseling intervention (condition #1) after completing the week 26 assessment. The primary trial outcome will be the change in internalized stigma from baseline to week 12 (following the most intensive part of the intervention). Change in internalized stigma from baseline to week 26 will be a secondary outcome to determine lasting effects of the intervention in a "maintenance" period with less frequent intervention. Other secondary outcomes will include depression, anxiety, stress, coping, and health-related quality of life (HRQOL)

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* At least one of the following stigmatized health conditions:
* Obesity (or high body weight that negatively affects health)
* Skin disease (including but not limited to psoriasis, eczema, or vitiligo)
* Cancer (including but not limited to lung, breast, cervical, colorectal, gynecologic, prostate, or head and neck; including individuals in remission)
* HIV
* Type 1 or type 2 diabetes
* Chronic pain
* Reported internalization of health-related stigma, as determined by a pre-specified cutoff score on internalized stigma measure and confirmed by interview

Participants must have availability to attend weekly virtual group meetings for 12 weeks, followed by every-other-week and monthly meetings through 26 weeks, in the evening on a specified weekday. Participants must be willing to actively participate and share information about themselves in the group meetings.

Participants must be able to read, comprehend, and speak English in order to participate in group sessions and complete study questionnaires.

Participation requires an electronic device (computer, tablet, or phone) with video capabilities and internet, wi-fi, or cellular data in order to attend group sessions and complete study questionnaires. Individuals who do not have such devices or internet access will still be eligible to participate. In such cases, screening procedures will be conducted by phone, and randomized participants will be provided with web cameras or internet-enabled devices (and/or provided with pre-paid cellular data) to facilitate participation.

Exclusion Criteria:

* Current or recent (e.g., past 3 months) receipt of psychotherapy or a psychosocial or peer support intervention (exceptions may be made if therapy or support is not focused on health conditions and is unlikely to affect internalized health-related stigma; e.g., family or marriage counseling, religious study groups, etc.)
* Psychiatric hospitalization in the past 6 months
* Recent (e.g., past 3 months, approximately) change in medications taken for psychiatric reasons
* Current, active suicidal thoughts or suicide attempt within the past year
* Current or past thought disorder or psychosis, or unmanaged bipolar disorder
* Current alcohol/substance use disorder that requires immediate treatment
* Health-related stigma due primarily to mental illness or substance use, or due to health conditions not specified in inclusion criteria.
* No reported internalization of health-related stigma and/or score below pre-specified cutoff on internalized stigma measure
* Unwilling or unable to complete study procedures

Participants with severe progression of disease (e.g., end-of-life) or who are undergoing acute, intensive treatment (such as chemotherapy or radiation therapy) will not be eligible to participate due to expected impacts on HRQOL and greater needs for psychological support than the intervention is intended to provide. Such participants may be eligible after completion of acute treatment or if severe symptoms remit and/or prognosis improves.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Estimated)
Dates: Start 2024-10-03 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in Internalized Health-Related Stigma Scale score at Week 12 | Baseline to Week 12
  Estimated mean change score for the total scale (primary outcome) and three subscales (Perceived and Anticipated Stigma, Stereotype Application and Self-Devaluation, and Stigma Resistance); scale scores are averaged and range from 1-7, with higher scores indicating greater internalized health-related stigma.

SECONDARY OUTCOMES:
Change in Internalized Health-Related Stigma Scale score at Week 26 | Baseline to Week 26
  Estimated mean change score for the total scale (primary outcome) and three subscales (Perceived and Anticipated Stigma, Stereotype Application and Self-Devaluation, and Stigma Resistance); scale scores are averaged and range from 1-7, with higher scores indicating greater internalized health-related stigma.
Change in Internalized Shame Scale score at Week 12 | Baseline to Week 12
  Estimated mean change score for two subscales: Shame (summed scores range from 0-96, higher scores indicate greater shame) and Self-Esteem (summed scores range from 0-24, higher scores indicate higher self-esteem).
Change in Internalized Shame Scale score at Week 26 | Baseline to Week 26
  Estimated mean change score for two subscales: Shame (summed scores range from 0-96, higher scores indicate greater shame) and Self-Esteem (summed scores range from 0-24, higher scores indicate higher self-esteem).
Change in UCLA Loneliness Scale score at Week 12 | Baseline to Week 12
  Estimated mean change score, with summed scores ranging from 20-80 (higher scores indicate greater loneliness/isolation).
Change in UCLA Loneliness Scale score at Week 26 | Baseline to Week 26
  Estimated mean change score, with summed scores ranging from 20-80 (higher scores indicate greater loneliness/isolation).
Change in Patient Health Questionnaire-9 score at Week 12 | Baseline to Week 12
  Estimated mean change score, with summed scores ranging from 0-27 (higher scores indicate greater severity of depression symptoms).
Change in Patient Health Questionnaire-9 score at Week 26 | Baseline to Week 26
  Estimated mean change score, with summed scores ranging from 0-27 (higher scores indicate greater severity of depression symptoms).
Change in Generalized Anxiety Disorder-7 Questionnaire score at Week 12 | Baseline to Week 12
  Estimated mean change score, with summed scores ranging from 0-21 (higher scores indicate greater severity of generalized anxiety).
Change in Generalized Anxiety Disorder-7 Questionnaire score at Week 26 | Baseline to Week 26
  Estimated mean change score, with summed scores ranging from 0-21 (higher scores indicate greater severity of generalized anxiety).
Change in Severity Measure for Social Anxiety Disorder score at Week 12 | Baseline to Week 12
  Estimated mean change score, with summed scores ranging from 0-40 (higher scores indicate greater severity of social anxiety).
Change in Severity Measure for Social Anxiety Disorder score at Week 26 | Baseline to Week 26
  Estimated mean change score, with summed scores ranging from 0-40 (higher scores indicate greater severity of social anxiety).
Change in 4-item Perceived Stress Scale score at Week 12 | Baseline to Week 12
  Estimated mean change score, with summed scores ranging from 0-16 (higher scores indicate greater perceived stress).
Change in 4-item Perceived Stress Scale score at Week 26 | Baseline to Week 26
  Estimated mean change score, with summed scores ranging from 0-16 (higher scores indicate greater perceived stress).
Change in General Self-Efficacy Scale score at Week 12 | Baseline to Week 12
  Estimated mean change score, with summed scores ranging from 10-40 (higher scores indicate greater self-efficacy).
Change in General Self-Efficacy Scale score at Week 26 | Baseline to Week 26
  Estimated mean change score, with summed scores ranging from 10-40 (higher scores indicate greater self-efficacy).
Change in Revised Illness Perceptions Questionnaire scores at Week 12 | Baseline to Week 12
  Estimated mean change scores on four subscales: Consequences, Personal Control, Illness Coherence, and Emotional Representations. Scores for each subscale are averaged, with ratings ranging from 1-5, and higher scores Indicating greater perceived consequences, control, understanding, and emotional impacts of health conditions, respectively.
Change in Revised Illness Perceptions Questionnaire scores at Week 26 | Baseline to Week 26
  Estimated mean change scores on four subscales: Consequences, Personal Control, Illness Coherence, and Emotional Representations. Scores for each subscale are averaged, with ratings ranging from 1-5, and higher scores Indicating greater perceived consequences, control, understanding, and emotional impacts of health conditions, respectively.
Change in SF-12v2 scores at Week 12 | Baseline to Week 12
  Estimated mean change scores in mental and physical health component t-scores, with a population mean score of 50 and standard deviation of 10 (higher scores indicate better mental and physical health-related quality of life, respectively).
Change in SF-12v2 scores at Week 26 | Baseline to Week 26
  Estimated mean change scores in mental and physical health component t-scores, with a population mean score of 50 and standard deviation of 10 (higher scores indicate better mental and physical health-related quality of life, respectively).
Change in CDC Healthy Days Core Measure at Week 12 | Baseline to Week 12
  Estimated mean change scores in items assessing the number of unhealthy days due to physical and mental health, respectively (range 0-30 days), the number of days of impairment due to poor health (0-30 days), and an unhealthy days index score of total combined physically and mentally unhealthy days (0-30 days).
Change in CDC Healthy Days Core Measure at Week 26 | Baseline to Week 26
  Estimated mean change scores in items assessing the number of unhealthy days due to physical and mental health, respectively (range 0-30 days), the number of days of impairment due to poor health (0-30 days), and an unhealthy days index score of total combined physically and mentally unhealthy days (0-30 days).

OTHER OUTCOMES:
Change in Brief COPE scores at Week 12 | Baseline to Week 12
  Estimated mean change in scores on the following subscales (all with two items rated 1-4, summed to produce scores ranging from 2-8, with higher scores indicating greater use of the respective coping strategy): self-distraction; active coping; denial; substance use; use of emotional support; use of instrumental support; behavioral disengagement; venting; positive reframing; planning; humor; acceptance; religion; and self-blame. Coping strategies may also be analyzed by grouping coping strategies into three broad categories and averaging scores for items within each category: active coping (active coping, positive reframing, planning, humor, acceptance); disengaged coping (self-distraction, denial, substance use, behavioral disengagement, venting, self-blame); and support coping (emotional support, instrumental support, religion).
Change in Brief COPE scores at Week 26 | Baseline to Week 26
  Estimated mean change in scores on the following subscales (all with two items rated 1-4, summed to produce scores ranging from 2-8, with higher scores indicating greater use of the respective coping strategy): self-distraction; active coping; denial; substance use; use of emotional support; use of instrumental support; behavioral disengagement; venting; positive reframing; planning; humor; acceptance; religion; and self-blame. Coping strategies may also be analyzed by grouping coping strategies into three broad categories and averaging scores for items within each category: active coping (active coping, positive reframing, planning, humor, acceptance); disengaged coping (self-distraction, denial, substance use, behavioral disengagement, venting, self-blame); and support coping (emotional support, instrumental support, religion).
Change in 6-Item Social Support Questionnaire scores at Week 12 | Baseline to Week 12
  Estimated mean change scores on two subscales assessing (1) the average number of support persons (N subscale) and (2) the average level of satisfaction with social support (the S subscale, with scores ranging from 1-6, and higher scores indicating greater satisfaction with social support).
Change in 6-Item Social Support Questionnaire scores at Week 26 | Baseline to Week 26
  Estimated mean change scores on two subscales assessing (1) the average number of support persons (N subscale) and (2) the average level of satisfaction with social support (the S subscale, with scores ranging from 1-6, and higher scores indicating greater satisfaction with social support).
Treatment Acceptability ratings at Week 12 | Week 12
  To assess treatment acceptability, participants in the two active treatment groups (not the waitlist control group) rate from 1-7 how acceptable and helpful the program was, how much they liked the program, and how satisfied they were; scores for these 4 items are averaged. Participants also rate (1-7) how likely they would be to recommend the program to others and the extent to which they learned new things, changed their attitudes about themselves, and the program helped with managing their health conditions. Participants also rate how much they learned and used specific skills from the program; these item responses are averaged on a 1-7 scale for learned skills and on a 1-5 scale for used skills. Higher scores indicate greater treatment acceptability.
Treatment Acceptability ratings at Week 26 | Week 26
  To assess treatment acceptability, participants in the two active treatment groups (not the waitlist control group) rate from 1-7 how acceptable and helpful the program was, how much they liked the program, and how satisfied they were; scores for these 4 items are averaged. Participants also rate (1-7) how likely they would be to recommend the program to others and the extent to which they learned new things, changed their attitudes about themselves, and the program helped with managing their health conditions. Participants also rate how much they learned and used specific skills from the program; these item responses are averaged on a 1-7 scale for learned skills and on a 1-5 scale for used skills. Higher scores indicate greater treatment acceptability.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Pearl, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared via the National Institute of Mental Health (NIMH) Data Archive (NDA; https://nda.nih.gov).
Supporting Information: Study Protocol, SAP
Time Frame: Data will be deposited to NDA starting 12 months after the award begins and will be deposited every six months thereafter following the usual NDA data submission dates of January 15th and July 15th.